CLINICAL TRIAL: NCT01619072
Title: A Randomized Controlled Community Study of the Effectiveness of Misoprostol for PPH Treatment at the Community Level (Home Births Attended by Primary Care Unit Staff) in Etay El Barood and Kafr El Dawar Districts (El Beheira Governorate), Egypt
Brief Title: Misoprostol for Treatment of Postpartum Hemorrhage at Community-level Births in Egypt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: Ministry of Health and Population, Egypt (Other Government); El Galaa Teaching Hospital (Other); Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3001
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Postpartum Hemorrhage
Keywords: postpartum hemorrhage; treatment; misoprostol; home births
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol; Referral and Consultation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Misoprostol (Active Comparator): 800 mcg sublingual misoprostol + referral to higher level care
  Interventions: Other: Misoprostol + referral
- Placebo (Placebo Comparator): Placebo + referral to higher level care
  Interventions: Other: Placebo + referral

INTERVENTIONS:
Other: Misoprostol + referral — 800 mcg of sublingual misoprostol (four tablets of 200 mcg misoprostol) + standard of care (referral to higher level care)
  Arms: Misoprostol
Other: Placebo + referral — Placebo (4 tablets resembling misoprostol) + standard of care (referral to higher level care)
  Arms: Placebo

SUMMARY:
This randomized controlled community-based trial will assess the effectiveness of administration of 800 mcg sublingual misoprostol with standard of care vs. placebo with standard of care for postpartum hemorrhage treatment at the community level, primarily home births attended by primary health care unit (PHU) staff in Etay El Barood and Kafr El Dawar districts (El Beheira governorate), Egypt. Standard of care per national guidelines in this setting is referral to a higher level health facility.

DETAILED DESCRIPTION:
Hospital-based clinical trials have demonstrated misoprostol to be a safe and effective treatment option for postpartum hemorrhage (PPH). Additional research is needed to demonstrate how these findings translate into program effectiveness at lower levels of the health care system, including community home births, where access to skilled providers and treatment options are limited and misoprostol could potentially have the greatest impact on maternal health outcomes. This randomized controlled community treatment trial will assess the effectiveness of misoprostol with standard of care (i.e., referral to higher level care) vs. placebo with standard of care for PPH treatment at the community level, primarily home births attended by primary health care unit staff in Etay El Barood and Kafr El Dawar districts (El Beheira governorate), Egypt. This research will help guide decisions on how to introduce misoprostol into PPH care programs in different contexts such as primary care settings, including community-based home births.

ELIGIBILITY:
Inclusion Criteria:

* women delivering with provider from participating primary health unit (PHU)
* willing and able to give informed consent
* vaginal delivery

Exclusion Criteria:

* women too advanced into active labor to provide informed consent
* known allergy to misoprostol and/or other prostaglandin
* women presenting with pregnancy complications, such as hypertension, suspected multiple pregnancy, previous caesarean section, suspected still birth, antepartum hemorrhage, previous complication in the third trimester (should be referred to higher level care for delivery)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2012-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin measurement of >2 g/dL pre- to -post-delivery. | Before delivery (at onset of labor), after delivery (2 to 4 days after delivery)
  Proportion of women with a change in hemoglobin of >2 g/dL pre- to post-delivery, as measured by the HemoCue machine at both time points.

SECONDARY OUTCOMES:
Proportion of women transferred to higher level care | Within 2 to 4 days after delivery
  Proportion of women transferred to higher level care will be compared. The condition of the woman at time of transfer and arrival will also be noted.
Proportion of women receiving additional interventions to treat PPH | Within 2 to 4 days after delivery
  Proportion of women who receive any additional intervention (e.g. uterotonics, manual removal of placental fragments, bimanual compression, IV fluids given, surgical procedures, blood transfusion, etc.) provided either at deliver site or upon transfer to district hospital.
Proportion of women with side effects | Within 24 hours of delivery
  Proportion of women with observed side effects (including shivering/chills, fever, nausea, diarrhea or fainting). Reported severity of side effects (classified by provider as "mild, "moderate," "severe," ), duration of side effects and proportion of of women receiving additional care to manage side effects will also be assessed.
Cost-effectiveness | Within 2 to 4 days after delivery
  A cost-effectiveness analysis will be done to compare the two treatment arms. The analysis will factor in the cost of materials used, procedures/interventions performed, transfers, and training of providers.
Proportion of women for whom intervention was correctly administered | Within 1 hour of PPH diagnosis
  Proportion of women for whom treatment was administered as described in protocol (referral initiated and tablets administered to woman after PPH diagnosis made)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Cherine Ramadan, MD, Principal Investigator — El Galaa Teaching Hospital; Nevine Hassanein, MD, Principal Investigator — Consultant; Emad Darwish, MD, Principal Investigator — Alexandria University Faculy of Medicine; Emad Ezzat, MD, Principal Investigator — Ministry of health and population; Rasha Dabash, MPH, Principal Investigator — Gynuity Health Projects
Locations (1):
- Prinary Health Units, Etay El Barood and Kafr El Dawar Districts, Beheira, Egypt

REFERENCES:
- [Derived] Parry Smith WR, Papadopoulou A, Thomas E, Tobias A, Price MJ, Meher S, Alfirevic Z, Weeks AD, Hofmeyr GJ, Gulmezoglu AM, Widmer M, Oladapo OT, Vogel JP, Althabe F, Coomarasamy A, Gallos ID. Uterotonic agents for first-line treatment of postpartum haemorrhage: a network meta-analysis. Cochrane Database Syst Rev. 2020 Nov 24;11(11):CD012754. doi: 10.1002/14651858.CD012754.pub2. PMID 33232518
- See also: Related Info — http://www.gynuity.org